CLINICAL TRIAL: NCT00513890
Title: Interest of Non Invasive Ventilation Versus Oxygen During the Intial Managment of Infant With Bronchiolitis Who Didn't Require Mechanical Ventilation
Brief Title: Interest of Non Invasive Ventilation Versus Oxygen During the Intial Managment of Infant With Bronchiolitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UF 7873
Record Dates: First submitted 2007-08-08; First posted 2007-08-09 (Estimated); Last update posted 2013-10-24 (Estimated); Status verified 2012-04

CONDITIONS: Bronchiolitis; Respiratory Distress
Keywords: Bronchiolitis; Esophageal pressure mesurement; Clinical score; Citical care; Infant
MeSH Terms: conditions — Bronchiolitis; Dyspnea

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Infantflow [EME, Brighton, England]

SUMMARY:
The purpose of the study is to evaluate, in a prospective way, the clinical, the manometric an gazometric benefit of non-invasive ventilation (VNI), (INFANTFLOW [EME, Brighton, England]) during bronchiolitis of the infant compared to a conventional managment.

DETAILED DESCRIPTION:
1. Experimental plan: The infants (0 to 6 month) admitted in pediatric intesive care unit for respiratory distress with bronchiolitis but not requiring mechanical ventilation are randomized in two groups: group "A" is treated with a non-invasive ventilation device(Infantflow) during 6 hours, group "B" is treated conventionally by inhalation of a Air/O2 mixture during 6 hours.
2. Outcome: Primary outcome: clinical score of respiratory distress at H0 and H6. Secondary outcome: respiratory and cardiac frequency, average blood pressure. Manometric: Variation of esophageal pressure at H0, H6. Gasometric: Minimal FiO2 necessary to reach an oxygen saturation between 94 and 98%, transcutaneus PCO2, PaO2/FiO2
3. Analyze results: Intention to treat analysis after having checked the randomization by comparing clinical gravity in the two arms (clinical score).
4. Calendar of the study: October 2006 at April 2008
5. Follow-up of the patients: the study proceeds during the hospitalization of the infants during 6 hours and will not impose any specific follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Infant from 0 to 6 months admitted in the PICU
* Clinical diagnosis: bronchiolitis
* Signs of respiratory distress evaluated with a clinical score of respiratory distress > 4

Exclusion Criteria:

* Cardiopathy, cystic fibrosis or a neuromuscular desease
* Need for mechanical ventilation

Ages: 1 Day to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 19 (Actual)
Dates: Start 2006-10; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Clinical score of respiratory distress at base line (H0) and at 6 hours (H6)
after the begining of the procedure.
The respiratory distress was evaluated with the modified Woods Clinical Asthma
Score (m-WCAS) [Hollman G, Shen G, Zeng L, et al. Crit Care Med 1998; 26:1731-1736]

SECONDARY OUTCOMES:
Clinical items: respiratory and cardiac rate, average blood pressure at H0 and H6.
Manometric: Variation of esophageal pressure at H0 and H6.
Gasometric: Minimal FiO2 necessary to reach an oxygen saturation between 94
and 98%, transcutanée PCO2, PaO2/FiO2

CONTACTS AND LOCATIONS:
Overall Officials: PICAUD Jean Charles, Doctor, Principal Investigator — Service de réanimation pédiatrique
Locations (1):
- Service réanimation Pédiatrique, Montpellier, Languedoc-Roussillon, France